CLINICAL TRIAL: NCT04506216
Title: Prevalence of Eating Disorders in Adult Patients With Type I Diabetes and Insulin Pump Treatment
Brief Title: Eating Disorders in Type 1 Insulin-dependent Diabetes Patients
Acronym: Diaboulimia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icadom (Industry)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A00147-32
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes; Eating Disorders
Keywords: diaboulimia; insulin pump treatment; DT1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders | interventions — Cohort Studies

STUDY DESIGN:
Intervention Model Description: cohort prospective monocentric
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort (Experimental): adult patients with type 1 diabetes and insulin pump treatment . Duration of participation: 30 minutes
  Interventions: Other: cohort

INTERVENTIONS:
Other: cohort — During a regular follow-up visit, the following data will be collected:
  * questionnaires on lifestyle, eating custom (SCOFF-F, 5th question of the m-SCOFF) and physical activity (IPAQ)
  * bio-electric impedance analysis
  * insulin pump and sensor data collection

SUMMARY:
The purpose of this study is to determine the prevalence of eating disorders in type 1 insulin-dependent diabetes patients

DETAILED DESCRIPTION:
The risk of developing an eating disorder is increased in type 1 diabetes patients and associated with a poor prognosis in terms of glycemic control, metabolic complications, degenerative complications, and mortality.

Therefore the terminology diaboulimia has emerged to characterize an eating disorder specific to type 1 insulin-dependent diabetes patients, with insulin under dosage with a view of losing or controlling weight and that can contribute to a deterioration of the body composition.

The purpose of this study is to determine the prevalence of eating disorders in an adult cohort with type 1 insulin-dependent diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age with type 1 diabetes treated with a subcutaneous insulin pump
* Patient followed up for a subcutaneous insulin pump treatment by the healthcare provider, participating in the study (Agir à Dom group).
* Beneficiary of social security coverage.

Exclusion Criteria:

* Patient with type 2 diabetes or MODY diabetes
* Patient wearing a pacemaker
* Breastfeeding or pregnant woman
* Deprived of liberty by judicial or administrative decision
* Legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Eating disorders in men and women | at inclusion
  To determine eating disorder prevalence in differentiated adult men and women with type 1 insulin-dependent diabetes.
  Patients answer to the SCOFF-F questions :
  * do you make yourself sick because you feel uncomfortably full?
  * do you worry that you have lost control over how much you eat?
  * have you recently lost more than one stone in a 3 month period?
  * do you believe yourself to be fat when others say you are too thin?
  * would you say that food dominates your life?
  Every "yes" attributes one point and gives a final score between 0 and 5; a score ≥2 indicates an eating disorder.

SECONDARY OUTCOMES:
Eating disorders in cohort | at inclusion
  To determine eating disorder prevalence in undifferentiated cohort (men and woman) with type 1 insulin-dependent diabetes.
  Patients answer to the SCOFF-F questions :
  * do you make yourself sick because you feel uncomfortably full?
  * do you worry that you have lost control over how much you eat?
  * have you recently lost more than one stone in a 3 month period?
  * do you believe yourself to be fat when others say you are too thin?
  * would you say that food dominates your life?
  Every "yes" attributes one point and gives a final score between 0 and 5; a score ≥2 indicates an eating disorder.
Auto declared insulin under dosage | at inclusion
  To Determine the auto declared insulin under dosage prevalence in undifferentiated cohort (men and woman) with type 1 insulin-dependent diabetes.
  Patients answer to the 5th m-SCOFF question :
  - do you ever take less insulin than you should?
  A "yes" answer means that patient underdoses insulin treatment.
Overall glycemia | at inclusion
  To identify if there is a link between an eating disorder and overall glycemic control, we will look after the last biological value of HbA1c rates
Basal/Bolus insulin ratio | at inclusion
  To identify if there is a link between an eating disorder and basal/bolus insulin ratio, we will extract and compare to eating disorder presence, this daily data from insulin pump over the 14 days preceding inclusion
Boluses performed per day | at inclusion
  To identify if there is a link between an eating disorder and boluses performed per day, we will extract and compare to eating disorder presence, this daily data from insulin pump over the 14 days preceding inclusion
Body composition | at inclusion
  To identify if there is a link between an eating disorder and body composition, we will perform a bio-electric impedance analysis and compare the result to eating disorder presence.
Continuous glycemic control | at inclusion
  To identify if there is a link between an eating disorder and continuous glycemic control, we will extract and compare to eating disorder presence, this data from the continuous glucose monitoring system (CGMS) over the 14 days preceding inclusion Glycemic control will be determined by the percentage of daily time into the glycemic target (between 70 and 180 mg/dL).
Glycemic variability | at inclusion
  To identify if there is a link between an eating disorder and glycemic variability, we will extract and compare to eating disorder presence, this data from the continuous glucose monitoring system (CGMS) over the 14 days preceding inclusion Glycemic variability will be determined by the Mean Amplitude of Glycemic Excursions (MAGE) algorithm.
Adherence to the sensor | at inclusion
  To identify if there is a link between an eating disorder and the adherence to the continuous glucose monitoring system (CGMS), we will extract and compare to eating disorder presence, this data from the continuous glucose monitoring system (CGMS) over the 14 days preceding inclusion Adherence will be determined by the number of minutes worn per day.
Blood glucose monitoring | at inclusion
  To identify if there is a link between an eating disorder and blood glucose monitoring, we will extract and compare to eating disorder presence, this data from the continuous glucose monitoring system (CGMS) over the 14 days preceding inclusion The monitoring will be determined by the number of scans done per day.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Bétry, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- AGIR à dom., Meylan, France

IPD SHARING:
Plan to Share IPD: Yes
Contact icadom@agiradom.com for any data request. The researcher will be invited to complete a form (data sharing agreement) explaining the reasons and the aim of the data requests. The data will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2022 to January 2037
Access Criteria: Researchers requesting the data have to be able to present a scientific reason to get access